CLINICAL TRIAL: NCT06447558
Title: The Effects of "Oral Administration of Breast Milk Droplets" and "Palatal Stimulation With a Finger" Methods on Feed Tolerance in Preterm Newborns Fed Via an Orogastric Tube
Brief Title: The Effects of "Oral Administration of Breast Milk Droplets" and "Palatal Stimulation With a Finger"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, aysel kokcudogan, Assistant professor, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: E-10840098-772.02-4979
Record Dates: First submitted 2024-04-20; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Infants
Keywords: Breast milk; Palatal stimulation with a finger

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Breast milk droplets group (No Intervention): We fed the infants via OGT in the oral administration of breast milk droplets group after applying a total of 0.5 cc of breast milk in drops into their mouths for 5 minutes by using an insulin injector.Breast milk droplets group was 30 infants
- Palatal stimulation group (Other): In the palatal stimulation group, following the necessary hygiene rules, we used the little finger of one of our hands with a glove on and stimulated the palate and gums of the infants with this finger by slow and peristalsis-like movements for 5 minutes while the infants were fed via OGT. Palatal stimulation group was 30 infants.
  Interventions: Behavioral: palatal stimulation with a finger in premature infants
- Control group (No Intervention): We fed the premature infants in the control group via OGT following all hygiene rules, but we performed no intervention. In the intervention groups, where we orally applied breast milk in droplets in one group and stimulated the palate of the newborns by using a finger in the other, we performed these interventions every 3 hours for 5 minutes for 7 days at feeding times.

INTERVENTIONS:
Behavioral: palatal stimulation with a finger in premature infants — Oral administration of breast milk droplets, palatal stimulation with a finger in premature infants
  Arms: Palatal stimulation group

SUMMARY:
The aim of this study was to investigate the effects of "oral administration of breast milk droplets" and "finger palatal stimulation" on feeding tolerance in preterm neonates fed with orogastric tube feeding.

This randomized controlled experimental study was conducted in the neonatal intensive care unit of a private hospital. The study included 90 premature newborns born at 28-36 weeks of gestation and admitted to the intensive care unit. The intervention group consisted of 60 infants and the control group consisted of 30 infants. "Demographic Information Form" and "Patient Follow-up Form" were used to collect data. Data collection tools were used before, during and after the procedures in all groups. In one of the intervention groups, breast milk droplets were applied to the oral cavity of the newborns, and in the other group, the palate of the newborns was stimulated using a finger. These interventions were performed for 5 minutes every 3 hours for 7 days during the newborns' feeding times. Neonates in the control group were fed with an orogastric tube by following hygiene rules, but no study intervention was performed in these infants. SPSS (Statistical Package for Social Sciences) 22.0 for Windows software was used for statistical analysis.

DETAILED DESCRIPTION:
This is a randomized, controlled and experimental study investigating the effects of "oral administration of breast milk droplets" and "finger palatal stimulation" methods on feeding tolerance in infants fed with an orogastric tube.The study included 90 premature infants who were 28-36 weeks of gestation, admitted to the neonatal intensive care unit and whose parents consented to participate. Two intervention groups (Intervention1 and Intervention2) consisted of a total of 60 infants and the control group consisted of 30 infants. A power analysis was conducted to calculate the number of premature infants to be included in the study. We created the randomization table using the instructions in the following link: "https://www.calculatorsoup". The study was completed with 90 newborns who met the inclusion criteria and whose parents consented to participate. Of these newborns, 60 were in the intervention group and 30 were in the control group. Data were collected using the "Demographic Information Form" and "Patient Follow-up Form" developed by the researcher in line with the literature.

Study Execution

Pre-Procedure: The steps before the procedure were the same for each group, i.e. the oral administration of breast milk droplets group, the palatal stimulation group and the control group. Before the procedure, the subjects' identities were checked and the Demographic Information Form (gender, gestational week, birth weight, head circumference and height) and Patient Follow-up Form were completed. The newborns in all groups were placed on an orogastric tube, positioned, and finally the infants' heads were gently lifted from the bed at a 30-degree angle. After achieving the correct position, their remains were checked and the results were noted. The stomachs of all premature infants included in the study were checked every 3 hours before feeding for 7 days.

Sequence of Procedures: Infants in the oral administration of breast milk droplets group were fed with an oroastric catheter after a total of 0.5 cc of breast milk was administered in drops using an insulin syringe for 5 minutes. In the palatal stimulation group, the palate and gums were stimulated with slow and peristalsis-like movements for 5 minutes with the gloved pinky finger of one hand while the infants were fed with an orogastric catheter, following the necessary hygiene rules. Premature infants in the control group were fed with orogastric catheter by following all hygiene rules, but no intervention was performed. Intervention groups received intervention for 5 minutes every 3 hours during feeding hours for 7 days.

Post Procedure: After feeding, all infants received routine comfort care, including diaper care, positioning, and environmental adjustments (adjusting sound and light levels, etc.). After routine comfort care, defecation was examined in all subjects every day during the 7-day follow-up period and the results were recorded. At the end of each day, the abdominal circumference and body weight of the newborns were measured and the measurements were noted on the forms. SPSS (Statistical Package for Social Sciences) 22.0 for Windows software was used for statistical analysis. Number, percentage, mean and standard deviation were used in descriptive statistical methods. Differences between the rates of categorical variables in independent groups were analyzed using the chi-square test and Fisher's exact test. One-way Analysis of Variance was used to compare quantitative continuous data between groups. Repeated Measures ANOVA Test was used for within-group comparisons.

ELIGIBILITY:
Inclusion Criteria:

* Babies born between 28-36 weeks of birth
* Premature babies without major congenital anomalies, severe systemic disorders, NEC, suspected or confirmed sepsis diagnosis
* Premature babies whose vital importance is fixed
* Babies who were not intubated at the time of the research

Exclusion Criteria:

* Babies younger than 28 weeks of birth and older than 36 weeks of birth
* Premature babies with major congenital anomalies, severe systemic disorders, NEC, suspected or confirmed sepsis diagnosis
* Premature babies whose vital features are unstable
* Babies who were intubated at the time of the research
* Babies who do not have parental permission to work

Ages: 28 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-06-28 (Actual)

PRIMARY OUTCOMES:
Defecation | 7 days
  The number of daily defecations was monitored
Residual control | 7 days
  Daily residue count was monitored
Body weight | 7 days
  Body weight checked daily
Abdominal circumference measurement | 7 days
  Abdominal circumference was measured daily

CONTACTS AND LOCATIONS:
Overall Officials: Aysel Kokcu Dogan, Study Chair — Medipol University
Locations (1):
- Medipol University, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No